CLINICAL TRIAL: NCT02445183
Title: COPDGene/Lung Cancer Center Database
Status: Completed | Type: Observational
Sponsor: National Jewish Health (Other)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: HS 2815
Record Dates: First submitted 2015-05-11; First posted 2015-05-15 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Lung Cancer; COPD
MeSH Terms: conditions — Lung Neoplasms; Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Lung Cancer: Confirmed diagnosis of lung cancer
  Interventions: Other: None, N/A
- No Lung Cancer Controls: Unconfirmed lung cancer diagnosis, false positive
  Interventions: Other: None, N/A

INTERVENTIONS:
Other: None, N/A

SUMMARY:
The COPDGene® / Lung Cancer Database Study is a nested case-control study. This study is an ancillary study to COPDGene® Phase 1 and Phase 2. Lung cancer cases, which have been reported by COPDGene® subjects since the time of COPDGene® study enrollment, will be retrospectively verified with additional medical data collection pertaining to lung cancer. Additional 'control' subjects will also be identified and verified as a 'no lung cancer controls'. Data previously collected through the COPDGene® Study, including QCT results and clinical results (medication use, rate of acute exacerbations of COPD, etc) will be used as variables for analysis.

DETAILED DESCRIPTION:
COPDGene® subjects will be screened through several mechanisms for enrollment into the Lung Cancer Database:

1. The COPDGene® Phase 1 Longitudinal Follow-up Questionnaire.
2. The COPDGene® Phase 2 Medical History Questionnaire at Visit 1
3. Medical Records Collection through the Mortality Adjudication Committee

Potential cases will be those who respond yes to lung cancer will be contacted by phone by a study coordinator and be screened for the COPDGene® Lung Cancer Database. Medical records will be analyzed to determine the patient's cancer diagnosis, pathology, and treatment. Information will be collected at each individual institution, de-identified, and entered into the password-protected COPDGene® DCC lung cancer database, through a web-based interface. The survival data will be obtained through review of medical records or the Social Security Death Index in conjunction with the COPDGene® mortality adjudication committee. For the nested case-control study, controls will be matched from the those subjects on COPDGene who answered 'No' to the longitudinal follow-up question "have you been diagnosed with lung cancer" as per COPDGene protocol.

Medical records regarding the patient's cancer diagnosis, pathology and treatment will be collected following signed release of medical information from the patient. The following information will be collected and entered into a database. The survival data will be obtained through review of medical records or the Social Security Death Index.

i. Date of diagnosis ii. Type of specimen iii. Laterality iv. Lobe v. Record of any false positives (can be used as verified controls) b. Pathology Findings: i. Histology ii. Molecular Analysis, if done. iii. Stage (TNM classification) iv. Histologic grade c. Treatment i. Surgery ii. Radiation iii. Chemotherapy iv. Presentation at Tumor Board d. Outcomes i. Recurrence, Second primary cancers ii. Survival after cancer diagnosis, Cause of death Study coordinators at each site contact subjects who have self-reported lung cancer or were identified as having lung cancer by follow-up clinic visits and complete the lung cancer data form. The data collected on each subject is de-identified at the recruiting site prior to being downloaded into the COPDGene® DCC located at National Jewish Health. A lung cancer adjudication committee, including Drs. Carr and Bowler, will review each case for accuracy and completeness.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet all of the following criteria

  1. Be enrolled in COPDGene® Phase 1 with or without enrollment in Phase 2 with newly diagnosed, (within the time of enrollment), non-small cell lung cancer (NSCLC) or small-cell lung cancer (SCLC).
  2. Documented GOLD stage 1-4 COPD or a history of smoking with no COPD
  3. Signed HIPAA Research Authorization and a Release of Protected Health Information form to collect and review medical records regarding lung cancer diagnosis, treatment, and outcome

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for study are those enrolled in the COPDGene®. Subjects will be screened for enrollment through the COPDGene® longitudinal follow-up questionnaire or during their Phase 2 visit. Those patients that answer yes to "since the last follow up have you been diagnosed with cancer?" will be contacted by a study coordinator and offered enrollment in the COPDGene®/Lung Cancer Database.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2013-12; Primary Completion 2020-09-22 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Identify lung cancer variables | 1.5 years
  Use existing COPDGene® quantitative HRCT and clinical data to perform a nested case-control study and perform a univariate analysis to select significant variables for the development of lung cancer.

SECONDARY OUTCOMES:
Probability of lung cancer based on variables | 1.5 years
  Construct a multivariate model from the results of the univariate analysis to calculate the odds ratios for the variables that predict lung cancer

CONTACTS AND LOCATIONS:
Locations (1):
- National Jewish Health, Denver, Colorado, United States

REFERENCES:
- [Derived] El Kaddouri B, Strand MJ, Baraghoshi D, Humphries SM, Charbonnier JP, van Rikxoort EM, Lynch DA. Fleischner Society Visual Emphysema CT Patterns Help Predict Progression of Emphysema in Current and Former Smokers: Results from the COPDGene Study. Radiology. 2021 Feb;298(2):441-449. doi: 10.1148/radiol.2020200563. Epub 2020 Dec 15. PMID 33320065
- [Derived] Bradford E, Jacobson S, Varasteh J, Comellas AP, Woodruff P, O'Neal W, DeMeo DL, Li X, Kim V, Cho M, Castaldi PJ, Hersh C, Silverman EK, Crapo JD, Kechris K, Bowler RP. The value of blood cytokines and chemokines in assessing COPD. Respir Res. 2017 Oct 24;18(1):180. doi: 10.1186/s12931-017-0662-2. PMID 29065892